CLINICAL TRIAL: NCT01226082
Title: The Effect of Transcranial Direct Current Stimulation for Chronic Pain on Ophthalmologic Parameters
Acronym: tDCS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Pain medicine unit, Tel aviv Sourasky medical center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TASMC-10-SB-411-CTIL
Record Dates: First submitted 2010-10-10; First posted 2010-10-21 (Estimated); Last update posted 2010-10-21 (Estimated); Status verified 2010-10

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Transcranial Direct Current Stimulation (Experimental)
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — Patients will recieve tDCS in a 5-day period of treatment
  Other Names: tDCS

SUMMARY:
tDCS is a noninvasive brain stimulation technique that utilizes low amplitude direct currents applied via scalp electrodes to modulate the level of cortical excitability.Several studies have demonstrated that tDCS applied over the sensory-motor cortex has been able to decrease pain sensation and to increase pain threshold in healthy subjects and in chronic pain patients. The aim of this study was to test whether daily sessions of anodal tDCS repeated for 5 consecutive days may be effective in reducing pain in a large number of chronic pain patients. The cathode is usually applied over the right forhead above the eye. The aim of the study is to test whether daily sessions of tDCS repeated for 5 consecutive days will influence on ophthalmologic parametrs.

DETAILED DESCRIPTION:
tDCS is a noninvasive brain stimulation technique that utilizes low amplitude direct currents applied via scalp electrodes to modulate the level of cortical excitability.Several studies have demonstrated that tDCS applied over the sensory-motor cortex has been able to decrease pain sensation and to increase pain threshold in healthy subjects and in chronic pain patients. The aim of this study was to test whether daily sessions of anodal tDCS repeated for 5 consecutive days may be effective in reducing pain in a large number of chronic pain patients. The cathode is usually applied over the right forhead above the eye. The aim of the study is to test whether daily sessions of tDCS repeated for 5 consecutive days will influence on ophthalmologic parametrs.

Patients will recieve tDCS in a 5-day period of treatment. The participants will go through full ophtalmologic examination before and after the treatmnet In addition to the ophtalmologic examination Pain will be measured using visual analog scale (VAS) for pain and the short form McGill questionnaire (SF-MPQ). Disability will be measured using the ( Pain Disability Index (PDI) of Life-54 scale (MSQoL-54). Depressive symptoms and anxiety will also be evaluated using the Center for Epidemiological Studies-Depression Scale and the State-trait Anxiety Inventory (STAI). Cognitive function will be mesured using minimental test.

ELIGIBILITY:
Inclusion Criteria:

* patients who suffer from chronic pain VAS>4

Exclusion Criteria:

* pregnancy
* scalp lacerations
* history of seizures
* metal implants in the head
* heart pace maker
* ophthalmologic disease.
* The presence of deep brain stimulation system

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-11 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Ophtalmologic examination parameters-visual acuity test, eye movement, field of vision, Tonometry (Intraocular Pressure Testing) | 5 days

SECONDARY OUTCOMES:
Pain relief | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Silviu Brill, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv Sourasky Medical Center, Pain Medicine Unit, Tel Aviv, Israel